CLINICAL TRIAL: NCT06603142
Title: A Multicenter, Randomized, Double-Blind, Parallel-Controlled Phase II/III Study to Evaluate the Efficacy and Safety of AR882 Capsules Compared to Febuxostat Tablets in Patients with Primary Gout and Hyperuricemia
Brief Title: Phase II/III Study of AR882 Capsules Compared to Febuxostat Tablets in Patients with Primary Gout and Hyperuricemia
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Guangzhou Ruianbo Pharmaceutical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APRAB-H001-P301
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Primary Gout; Hyperuricemia
Keywords: ULT; Gout; Hyperuricemia; URAT1
MeSH Terms: conditions — Hyperuricemia; Gout | interventions — Febuxostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AR882 50MG (Experimental): Titrated from 12.5 mg to 25 mg (2 weeks each), then 50 mg for 4 weeks, with matching Febuxostat placebo.
  Interventions: Drug: Febuxostat 20MG Placebo; Drug: AR882 25MG; Drug: AR882 12.5MG; Drug: Febuxostat 40MG Placebo
- Febuxostat 40MG (Active Comparator): Titrated from 20 mg (4 weeks) to 40 mg (4 weeks) Febuxostat, with matching AR882 placebo.
  Interventions: Drug: Febuxostat 20MG Tablets; Drug: AR882 25MG Placebo; Drug: AR882 12.5MG Placebo; Drug: Febuxostat 40MG Tablets
- AR882 75MG (Experimental): Titrated from 25 mg to 50 mg (2 weeks each), then 75 mg for 4 weeks, with matching Febuxostat placebo.
  Interventions: Drug: Febuxostat 20MG Placebo; Drug: AR882 25MG; Drug: Febuxostat 40MG Placebo

INTERVENTIONS:
Drug: Febuxostat 20MG Tablets — Febuxostat 20MG Tablets
  Arms: Febuxostat 40MG
Drug: Febuxostat 20MG Placebo — Febuxostat 20MG Placebo
  Arms: AR882 50MG; AR882 75MG
Drug: AR882 25MG — AR882 25 MG Capsules
  Arms: AR882 50MG; AR882 75MG
Drug: AR882 12.5MG — AR882 12.5 MG Capsules
  Arms: AR882 50MG
Drug: AR882 25MG Placebo — AR882 25MG Placebo
  Arms: Febuxostat 40MG
Drug: AR882 12.5MG Placebo — AR882 12.5MG Placebo
  Arms: Febuxostat 40MG
Drug: Febuxostat 40MG Tablets — Febuxostat 40MG Tablets
  Arms: Febuxostat 40MG
Drug: Febuxostat 40MG Placebo — Febuxostat 40MG Placebo
  Arms: AR882 50MG; AR882 75MG

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of AR882 Capsules in patients with primary gout and hyperuricemia. The main questions it aims to answer are:

What is the efficacy of AR882 Capsules in reducing serum uric acid levels in patients with primary gout and hyperuricemia?

Researchers will compare AR882 Capsules with Febuxostat Tablets to see :

Phase II: To explore the efficacy of AR882 Capsules in patients with primary gout and hyperuricemia, aiming to determine the dosing regimen for the Phase III study Phase III: To evaluate the efficacy of AR882 Capsules in patients with primary gout and hyperuricemia.

Participants will:

Be randomly assigned to receive either AR882 Capsules or Febuxostat Tablets. Undergo regular assessments of serum uric acid levels. Report any adverse events or side effects experienced during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 and ≤ 75 years of age at the time of signing the informed consent form (ICF)；
* History of gout according to the 2015 American College Rheumatology/European League Against Rheumatism (ACR/EULAR) Gout Classification Criteria，with serum urate (sUA) levels ≥480μmol/L；
* Body mass index (BMI) must be within the range of ≥ 18 to ≤ 35 kg/m2；
* Participants with childbearing potential must agree to use medically accepted effective contraception during the study period and for 3 months after the last dose
* Willing to participate in the study and sign the informed consent form.

Exclusion Criteria:

* Known or suspected allergy to the study drug or its components, or previous intolerance or contraindications to febuxostat；
* HbA1c ≥8% within 2 weeks prior to randomization；
* Any of the following laboratory test results within 2 weeks prior to randomization：WBC<3.0×109/L，Hb<90g/L，PLT<80×109/L，ASTorALT>1.5×ULN，TBIL>1.5×ULN，Scr>1.5×ULN，eGFR<60mL/min/1.73m2；
* Use of any other uric acid-lowering drugs or concomitant medications affecting uric acid levels (including but not limited to losartan, calcium channel blockers, fenofibrate, atorvastatin, α-glucosidase inhibitors, insulin sensitizers, DPP4 inhibitors, SGLT2 inhibitors, metformin) within 2 weeks prior to randomization, except for stable dose usage；
* Use of aspirin >100 mg/day or unstable dosage within 2 weeks prior to randomization；
* Use of any diuretics within 2 weeks prior to randomization；
* Use of a strong or moderate CYP2C9 inhibitor or BCRP substrate drugs (see Appendix 2) within 2 weeks prior to randomization；
* Secondary hyperuricemia due to tumors, chronic kidney disease, hematological diseases, medications, or hereditary hyperuricemia；
* Presence of unresolved gout attacks within 2 weeks prior to randomization；
* Imaging or clinical manifestations (e.g., hematuria, back pain) of kidney stones or urolithiasis within 2 weeks prior to randomization；
* Other joint lesions that may confound gouty arthritis, such as rheumatoid arthritis, septic arthritis, traumatic arthritis, psoriatic arthritis, pseudogout, systemic lupus erythematosus, or joint diseases caused by chemotherapy, radiotherapy, chronic lead poisoning, acute obstructive nephropathy, etc.;
* Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin and resected cervical intraepithelial neoplasia that has been successfully treated；
* Severe cardiovascular or cerebrovascular diseases, such as New York Heart Association (NYHA) Class III-IV congestive heart failure, uncontrolled hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg), QTcF interval (Fridericia's formula) prolongation (male >450 ms, female >470 ms), myocardial infarction, acute stroke, uncontrolled arrhythmia, or unstable angina within 12 months prior to screening；
* Unable to swallow oral medications or have gastrointestinal diseases that may interfere with drug absorption, or have active gastric or duodenal ulcers within 3 months prior to screening；
* Systemic diseases requiring immunosuppressive therapy, or vaccination within 2 weeks prior to randomization；
* Other severe or uncontrolled diseases；
* History of xanthinuria；
* Poor compliance (e.g., alcoholism, drug abuse) that may affect the safety and efficacy evaluation of the study drug, as judged by the investigator；
* Pregnant or breastfeeding women；
* Any acute inflammation or clinically significant active infection；
* Active hepatitis B (HBsAg positive and HBV-DNA >1000 IU/mL), or positive for serum HCV antibodies, HIV antibodies, or syphilis antibodies；
* Previous kidney removal and/or kidney transplantation；
* Major surgery within 3 months prior to randomization, or planned major surgery during the study；
* Blood donation (or blood loss) ≥400 mL or blood transfusion within 3 months prior to randomization；
* Participation in another drug clinical trial within 3 months prior to screening or within 5 half-lives of the investigational product (whichever is longer), or participation in a medical device clinical trial within 3 months prior to screening；
* Any other condition deemed unsuitable for study participation by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The percentage of participants with serum uric acid <360 μmol/L | 8 Weeks

SECONDARY OUTCOMES:
The percentage of participants with serum uric acid <300, 240 μmol/L | 8 Weeks
The percentage of participants with serum uric acid <360, 300, 240 μmol/L | 2, 4, and 6 Weeks
The absolute change in serum uric acid levels from baseline | 2, 4, 6, and 8 Weeks
The percentage change in serum uric acid levels from baseline | 2, 4, 6, and 8 Weeks
Serum uric acid levels | 2, 4, 6, and 8 Weeks
Adverse events | 8 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Science, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided